CLINICAL TRIAL: NCT04014062
Title: An Assessor-blind, Balanced, Randomized, Two-treatment, Two-period, Single-dose, Two-way, Crossover, Comparative, Pharmacokinetic and Pharmacodynamic Study of Subcutaneous Injections of INTP5 of Intas Pharmaceuticals Ltd., India Against Neulasta of Amgen Inc., USA in Healthy, Adult Human Subjects Under Fed Condition.
Brief Title: Comparative, Pharmacokinetic and Pharmacodynamic Study of Subcutaneous Injections of INTP5 of Intas Pharmaceuticals Ltd., India Against Neulasta of Amgen Inc., USA in Healthy, Adult Human Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intas Pharmaceuticals, Ltd. (Industry)
Collaborators: Lambda Therapeutic Research Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 0553-17
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Pharmacokinetic Bioequivalence Study in Human Healthy Volunteers
Keywords: Pegfilgrastim; Biosimilar; Bioequivalence; Pharmacokinetics; Pharmacodynamics; Safety; Healthy Volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study staff taking care of subject's safety and the laboratory personnel doing the sample analysis of pharmacokinetic, pharmacodynamic and immunogenicity data are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- INTP5 Period I Crossover (Experimental): Period I: Subjects received a single dose of INTP5 subcutaneously at a dose of 6 mg/0.6 mL.
  Period II: After the first treatment cycle and a six week wash out period, patients received a single dose of US Neulasta.
  Interventions: Combination Product: INTP5; Combination Product: US Neulasta
- US Neulasta Period I Crossover (Active Comparator): Period I: Subjects received a single dose US Neulasta subcutaneously at a dose of 6 mg/0.6 mL.
  Period II: After the first treatment cycle and a six week wash out period, patients received a single dose of INTP5.
  Interventions: Combination Product: INTP5; Combination Product: US Neulasta

INTERVENTIONS:
Combination Product: INTP5 — INTP5: A proposed pegfilgrastim biosimilar to US Neulasta.
Combination Product: US Neulasta — US Neulasta: FDA-approved pegfilgrastim innovator product.

SUMMARY:
The study was an assessor-blind, balanced, randomized, two-treatment, two-period, single-dose, two-way crossover, comparative, pharmacokinetic (PK) and pharmacodynamic (PD) study of subcutaneous (SC) Pegfilgrastim injection (6 mg/0.6 mL; INTP5 and US-Neulasta) in healthy, adult, human subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy adult human volunteers between 18 and 45 years of age (both inclusive) living in and around Ahmedabad city or western part of India.
2. Having body weight ≥50 kg and body mass index (BMI) between 18.5 and 29.9 (both inclusive), calculated as weight in kg/height in meter^2.
3. Not having any significant disease in medical history or clinically significant abnormal findings during screening, abdominal ultrasonography, medical history, clinical examination, laboratory evaluations, 12-lead ECG and chest X-ray (posterior-anterior view; within the last 6 months) recordings.
4. Volunteer who is a Non-smoker
5. Able to understand and comply with the study procedures, in the opinion of the investigator.
6. Able to give voluntary written informed consent for participation in the trial.
7. In case of female subjects:

   * Surgically sterilized at least 6 months prior to study participation;- Or - If a woman of childbearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.
   * Serum pregnancy test (for female subjects) must be negative.

Exclusion Criteria:

1. Known hypersensitivity to the study drug or its constituents and/or hypersensitivity to E. coli derived proteins, and/or previous exposure to the study drug.
2. History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
3. Known case of hereditary fructose intolerance.
4. Subjects with latex allergies will be excluded as the needle cover on the single-use pre-filled syringe contains dry natural rubber (latex).
5. Any clinically significant laboratory finding including ANC, platelet, RBC count or hemoglobin level at the time of screening.
6. Prior exposure to any peptide colony stimulating or growth factor, including erythropoietin, filgrastim or Pegfilgrastim; Prior exposure to vaccines, immunoglobulin preparations, or immunomodulator's within the past 6 months prior to receiving the first dose; evidence of E. coli diarrhea or diseases within 3 months.
7. Any history or presence of asthma (including aspirin-induced asthma) or nasal polyp or NSAIDs induced urticaria.
8. Subjects with a history of pulmonary infiltrate or pneumonia in the last 6 months.
9. History of any hematologic disease including sickle cell disorders.
10. Smokers, or who have smoked within last six months prior to start of the study.
11. Ingestion or use of any prescribed medication at any time within 1 month prior to receiving first dose in Period-I.
12. Receipt of over-the-counter medicines which have not yet cleared from the body (5 half-lives must have passed for the medicine to be considered to have cleared from the body).
13. A recent history of harmful use of alcohol, i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 mL of 40% distilled spirits, such as rum, whisky, brandy etc.) or consumption of alcohol or alcoholic products within 72 hours prior to receiving study medicine in Period-I.
14. Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.
15. Donation of blood (1 unit or 350 mL) or equivalent amount of blood substitute. Receipt of an investigational medicinal product or participation in a drug research study within a period of 180 days prior to the first dose of study medication. Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study.
16. Positive result for human immunodeficiency virus (HIV I &/or II) and/or hepatitis B and C tests.
17. History or presence of cancer because of which anticipated life span is less than 5 years as per the investigator's assessment.
18. History or presence of psychiatric disorders.
19. Presence of tattoo or scars or any type of skin lesions due to infection, burning, wound or inflammation at the proposed site of injection.
20. An unusual diet, for whatever reason (e.g. low-sodium), for 4 weeks prior to receiving the study medicine in Period-I. In any such case, subject selection will be at the discretion of the Principal Investigator.
21. Consumption of grape fruit or grape fruit products within 72 hours prior to receiving study drug in Period-I.
22. A history of difficulty in donating blood.
23. Females, pregnant or lactating, or planning to become pregnant during the course of the study or found positive in pregnancy test at screening.
24. Any infections in the last 4 weeks before receiving study medication in Period-I.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anshul Attrey, M.D., Principal Investigator — Lambda Therapeutic Research Ltd.; Vinu Jose, M.D., Study Director — Intas Pharmaceuticals, Ltd.
Locations (1):
- Lambda Therapeutic Research Ltd., Ahmedabad, Gota, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 144 subjects were planned and enrolled. Of these 144, 2 subjects withdrew before dosing. Hence, 142 subjects started the study, were dosed, and were considered for the study analyses.
Groups:
- INTP5 Period I, US Neulasta Period II Crossover: Period I: Subjects received a single dose of INTP5 subcutaneously at a dose of 6 mg/0.6 mL.
  Period II: After the first treatment cycle and a six week wash out period, patients received a single dose of US Neulasta.
  INTP5: INTP5: A proposed pegfilgrastim biosimilar to US Neulasta.
  US Neulasta: US Neulasta: FDA-approved pegfilgrastim innovator product.
- US Neulasta Period I, INTP5 Period II Crossover: Period I: Subjects received a single dose US Neulasta subcutaneously at a dose of 6 mg/0.6 mL.
  Period II: After the first treatment cycle and a six week wash out period, patients received a single dose of INTP5.
  INTP5: INTP5: A proposed pegfilgrastim biosimilar to US Neulasta.
  US Neulasta: US Neulasta: FDA-approved pegfilgrastim innovator product.
Period: Period I: Dosing
Arm/Group | INTP5 Period I, US Neulasta Period II Crossover | US Neulasta Period I, INTP5 Period II Crossover
Started | 71 | 71
Completed | 64 (Period I: Dosing, includes a washout period of 42 days before starting Period II: Crossover Dosing) | 65 (Period I: Dosing, includes a washout period of 42 days before starting Period II: Crossover Dosing)
Not Completed | 7 | 6
Not completed — Medical Grounds | 4 | 5
Not completed — Withdrawal by Subject | 3 | 1
Period: Period II: Crossover Dosing
Arm/Group | INTP5 Period I, US Neulasta Period II Crossover | US Neulasta Period I, INTP5 Period II Crossover
Started | 64 | 65
Completed | 64 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INTP5 Period I, US Neulasta Period II Crossover | US Neulasta Period I, INTP5 Period II Crossover | Total
Number analyzed (Participants) | 71 | 71 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (5.74) | 32.5 (6.38) | 33.6 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 36 | 72
  Male | 35 | 35 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 71 | 71 | 142
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 71 | 71 | 142
Height [Mean (Standard Deviation); unit: cm] | 159.1 (7.99) | 159.3 (9.00) | 159.2 (8.48)
Weight [Mean (Standard Deviation); unit: kg] | 60 (7.42) | 61.6 (8.49) | 60.8 (7.98)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.77 (2.788) | 24.32 (3.188) | 24.04 (2.996)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Endpoints: Pegfilgrastim C[Max]
Description: Maximum measured serum concentration, calculated from the serum concentration vs. time profile of the individual subjects.
Time Frame: Samples withdrawn at 1 hour pre-dose , at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 (D-2), 26, 30, 36, 42, 48 (D-3), 60, 72 (D-4), 96 (D-5), 120 (D-6), 144 (D-7), 168 (D-8), 192 (D-9), 240 (D-11), 288 (D-13), 336 (D-15) & 504 (D-22) hours post-dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- INTP5 Treatment: INTP5: A proposed pegfilgrastim biosimiar to US Neulasta. Outcomes Measures were grouped by treatment. This Group includes patients that received INTP5 in either Period I or Period II.
- US Neulasta Treatment: US Neulasta: FDA approved pegfilgrastim innovator product. Outcomes Measures were grouped by treatment. This Group includes patients that received US Neulasta in either Period I or Period II.
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 129 | 129
ng/mL | 474.269 (240.2247) | 425.578 (219.8054)

2. Primary Outcome: Pharmacokinetic (PK) Endpoints: Pegfilgrastim AUC[0-infinity]
Description: Area under the serum concentration versus time curve from time zero to infinity. Where AUC[0-infinity]= AUC[0-t] + Ct/λz(lambda-z), Ct is the last measurable concentration and λz(lambda-z) is the terminal rate constant.
Time Frame: as for outcome 1
Population: 3 subjects having three consecutive missing samples in the elimination phase were excluded from the statistical analysis of AUC0-t and other elimination phase dependent PK parameters
Measure: Mean (Standard Deviation); unit: ng.h/mL
Groups:
- INTP5 Treatment: INTP5: A proposed pegfilgrastim biosimilar to US Neulasta. Outcomes Measures were grouped by treatment. This Group includes patients that received INTP5 in either Period I or Period II.
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 128 | 127
ng.h/mL | 21015.8632 (12985.3760) | 18327.4192 (11156.1580)

3. Primary Outcome: Pharmacodynamic (PD) Endpoints: E[Max] for Baseline Non-adjusted ANC
Description: Maximum measured absolute neutrophil count (ANC).
Time Frame: Samples were withdrawn 1 hour pre-dose and at 6, 12, 24 (D-2), 36, 48 (D-3), 60, 72 (D-4), 96 (D-5), 120 (D-6), 144 (D-7), 168 (D-8), 192 (D-9), 216 (D-10), 240 (D-11), 288 (D-13), 312 (D-14), 336 (D-15), 360 (D-16) and 504 (D-22) hours post-dose.
Measure: Mean (Standard Deviation); unit: x10^3 cells/uL
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 129 | 129
x10^3 cells/uL | 38.82 (9.009) | 37.97 (9.258)

4. Primary Outcome: Pharmacodynamic (PD) Endpoints: AUEC[0-t] for Baseline Non-adjusted ANC
Description: Area under the absolute neutrophil count (ANC) versus time curve from time zero to the last measurable concentration as calculated by linear trapezoidal method.
Time Frame: as for outcome 3
Population: 5 subjects having three consecutive missing samples in the elimination phase were excluded from the statistical analysis of AUC0-t and other elimination phase dependent PD parameters.
Measure: Mean (Standard Deviation); unit: x10^3 cells*h/uL
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 128 | 125
x10^3 cells*h/uL | 6638.12 (1404.376) | 6554.04 (1465.072)

5. Secondary Outcome: PK Endpoint: Pegfilgrastim AUC[0-t]
Description: Area under the serum concentration vs. time curve, calculated by linear trapezoidal rule from measured data points from the time zero to the time of last quantified concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 128 | 127
ng.h/mL | 21001.567 (12983.9811) | 18312.112 (11156.5248)

6. Secondary Outcome: PK Endpoint: Pegfilgrastim T[Max]
Description: The time of observing the peak concentration, calculated from the serum concentration vs. time profile of the individual subjects.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 129 | 129
h | 26.189 (6.8110) | 25.754 (7.6188)

7. Secondary Outcome: PK Endpoint: Pegfilgrastim λz(Lambda-z)
Description: Terminal rate constant: First order rate constant associated with the terminal (log-linear) portion of the curve. This was estimated via linear regression of time vs. log concentration. This parameter was calculated by linear least squares regression analysis using last three or more nonzero plasma concentration values.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 128 | 127
1/h | 0.021 (0.0094) | 0.019 (0.0088)

8. Secondary Outcome: PK Endpoint: Pegfilgrastim R^2 Adjusted
Description: Goodness of fit statistic for the terminal phase, adjusted for the number of points used in the estimation of λz.
  R^2 is the coefficient of Determination and can range from 0 to 1,; with higher values indicating greater predictability.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Coefficient of Determination
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 128 | 127
Coefficient of Determination | 0.968 (0.0543) | 0.967 (0.0344)

9. Secondary Outcome: PK Endpoint: Pegfilgrastim t[1/2]
Description: The terminal half-life calculated using the formula 0.693/λz(lambda-z).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 129 | 129
h | 39.963 (18.5548) | 44.824 (29.3461)

10. Secondary Outcome: PK Endpoint: Pegfilgrastim AUC[_Percent_Extrap_Obs]
Description: The residual area in percentage determined by the formula, [(AUC[0-infinity]-AUC]0-t])/AUC0-infinity] x 100.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent of AUC
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 128 | 127
percent of AUC | 0.105 (0.117) | 0.139 (0.1726)

11. Secondary Outcome: PD Endpoint: T[Max] for Baseline Non-adjusted ANC
Description: Time to reach the maximum measured absolute neutrophil count (ANC)
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: h
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 129 | 129
h | 67.231 (16.0553) | 63.734 (13.1649)

12. Secondary Outcome: PD Endpoint: E[Max], Baseline-adjusted ANC
Description: Maximum measured absolute neutrophil count (ANC)
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: x10^3 cells/uL
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 129 | 129
x10^3 cells/uL | 34.66 (8.531) | 33.84 (8.863)

13. Secondary Outcome: PD Endpoint: AUEC[0-t], Baseline-adjusted ANC
Description: as for outcome 4
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: x10^3cells*h/uL
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 128 | 125
x10^3cells*h/uL | 4626.40 (1163.806) | 4565.80 (1278.987)

14. Secondary Outcome: PD Endpoint: T[Max], Baseline-adjusted ANC
Description: Time to reach the maximum measured absolute neutrophil count (ANC)
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: h
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 129 | 129
h | 67.231 (16.0553) | 63.734 (20.7)

15. Secondary Outcome: PD Endpoint: λz(Lamda-z) and Baseline-adjusted ANC
Description: First order rate constant associated with the terminal (log-linear) portion of the curve. This is estimated via linear regression of time vs. log concentration.
  This parameter will be calculated by linear least squares regression analysis using at least last three or more non-zero values.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 128 | 125
1/h | 0.02 (0.011) | 0.02 (0.013)

16. Secondary Outcome: PD Endpoint: t[1/2] for Baseline-adjusted ANC
Description: The terminal half-life will be calculated as 0.693/λz(lamda-z).
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 128 | 125
h | 55.98 (34.973) | 56.27 (31.671)

17. Other Pre Specified Outcome: Immunogenicity: Presence of Anti-drug Antibodies
Description: Evaluation of immunogenicity is carried out in a tiered fashion:
  1. Screening assay to assess if samples were positive or negative for anti-PegG-CSF.
  2. Confirmatory assays for samples that were positive in the screening assay. The confirmatory assays assessed if antibodies were specific for INTP5, Neulasta, PEG and/or filgrastim.
  3. Titer assay was performed to determine titer of the anti-PEG-GCSF antibody samples.
  4. Neutralizing antibody (NAb) assay for those samples that were positive in the confirmatory assays to assess the neutralizing capability of the antibody to inhibit pegfilgrastim activity.
Time Frame: 0-71 Days
Population: Only a fraction of the population was tested for Immunogenicity. Only participants that displayed treatment related AEs with plausible immune-mediated pathology were analysed for immunogenicity. The data below represents the outcomes for the fraction of each arm that was tested.
Measure: Count of Participants; unit: Participants
Groups:
- INTP5 Treatment: Period I: Subjects received a single dose of INTP5 subcutaneously at a dose of 6 mg/0.6 mL.
  Period II: After the first treatment cycle of US Neulasta and a six week wash out period, patients received a single dose of INTP5
  INTP5: A proposed pegfilgrastim biosimilar to US Neulasta. US Neulasta: FDA-approved pegfilgrastim innovator product.
- US Neulasta Treatment: Period I: Subjects received a single dose US Neulasta subcutaneously at a dose of 6 mg/0.6 mL.
  Period II: After the first treatment cycle of INTP5 and a six week wash out period, patients received a single dose of US Neulasta.
  INTP5: A proposed pegfilgrastim biosimilar to US Neulasta. US Neulasta: FDA-approved pegfilgrastim innovator product.
Arm/Group | INTP5 Treatment | US Neulasta Treatment
Number analyzed (Participants) | 64 | 65
Participants
  Period I: Negative for anti-drug- | 3 | 2
  Period I: Positive for anti-PegG-CSF | 1 | 1
  Period I: Not Tested for Immunogenicity | 60 | 62
  Period I: Neutralizing antibody | 0 | 0
  Period II: Negative for anti-drug- | 0 | 0
  Period II: Positive for anti-PegG-CSF | 0 | 0
  Period II: Not Tested for Immunogenicity | 64 | 65
  Period II: Neutralizing antibody | 0 | 0

ADVERSE EVENTS:
Time Frame: 79 days
Groups:
- INTP5 Treatment: INTP5: A proposed pegfilgrastim biosimiar to US Neulasta. Outcomes Measures were grouped by treatment. This Group includes patients that received INTP5 in either Period I or Period II.
  Given that this was a crossover design, AE totals for the entire study are reported comprehensively for Period I (71 Subjects) and Period II (65 Subjects) combined for the 136 subjects who received this treatment. Due to participant dropout between treatments, the number at risk for a given treatment is lower than the starting population for the study.
- US Neulasta Treatment: US Neulasta: FDA approved pegfilgrastim innovator product. Outcomes Measures were grouped by treatment. This Group includes patients that received US Neulasta in either Period I or Period II.
  Given that this was a crossover design, AE totals for the entire study are reported comprehensively for Period I (71 Subjects) and Period II (64 Subjects) combined for the 135 subjects who received this treatment. Due to participant dropout between treatments, the number at risk for a given treatment is lower than the starting population for the study.
Arm/Group | INTP5 Treatment | US Neulasta Treatment
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/135
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/135
Other Adverse Events (participants affected / at risk) | 39/136 | 39/135
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INTP5 Treatment (N=136) | US Neulasta Treatment (N=135)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Injection site pain (General disorders) | 2 (2) | 5 (5)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Human chorionic gonadotropin increased (Investigations) | 2 (2) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Red blood cells urine (Investigations) | 0 (0) | 1 (1)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 19 (19)
Headache (Nervous system disorders) | 12 (12) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-12-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT04014062/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT04014062/SAP_001.pdf